CLINICAL TRIAL: NCT06919913
Title: The Effect of Peri-Operative Adjunctive Probiotics on Immunological Markers in Cases of Prosthetic Joint Infection of the Hip and Knee
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-01249
Record Dates: First submitted 2025-03-27; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Prosthetic-joint Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic supplementation + Standard of care (Experimental): Patients will receive their first dose of the probiotic within 48 hours of starting post-operative antibiotic treatment. The probiotic is continued for the initial 6 weeks of antibiotic treatment in addition to standard of care (SOC).
  Interventions: Dietary Supplement: Culturelle Digestive Daily Probiotic Capsule
- Standard of care alone (No Intervention): Patients do not receive any additional treatment and undergo SOC treatment.

INTERVENTIONS:
Dietary Supplement: Culturelle Digestive Daily Probiotic Capsule — Each capsule contains 10 billion colony-forming units (CFU) of Lactobacillus rhamnosus GG. Subjects will self-administer 1 oral capsule daily for 6 weeks post operatively.
  Arms: Probiotic supplementation + Standard of care

SUMMARY:
The purpose of this study is to determine whether probiotics in addition to standard of care (SOC) can improve immunological markers following treatment for prosthetic joint infection (PJI). The study aims to determine whether probiotics in addition to SOC decrease immunological markers following treatment for PJI, improve medical and surgical complications and mortality in patients with PJI, and lead to improved gastrointestinal (GI)-specific patient reported outcomes measures (PROMs) in patients with PJI.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 18-90 years of age.
* Diagnosis of PJI based upon Musculoskeletal Infection Society (MSIS) criteria
* Planned treatment with surgical debridement, antibiotics, implant retention (DAIR), single- and two-stage revision total joint arthroplasty (TJA) for PJI with an anticipated plan for eventual discontinuation of oral/IV antibiotics.
* Patients with prior PJI in the same joint that has recurred.
* Patients who understand the benefits and risks associated with taking a probiotic and are willing and able to provide informed consent.

Exclusion Criteria:

* Fungal PJI.
* Inflammatory bowel disease, diverticulitis, history of intestinal surgery, or gastrointestinal issue where there is concern for gut integrity.
* Severe acute gastrointestinal diseases (active bowel leak, acute colitis, acute pancreatitis).
* Active endocarditis.
* History of pancreatitis
* History of intolerance to probiotics.
* Patients that are pregnant or lactating.
* Immunocompromised patients and patients with immunosuppressive conditions (uncontrolled HIV, chemotherapy for cancer treatment, stem cell transplantation, immunosuppressive medications for solid organ transplant, systematic corticosteroid use, immunosuppressive medications for autoimmune dysfunction, and neonates).
* Patients who are critically ill.
* Revision TJA for aseptic reasons.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in erythrocyte sedimentation rate (ESR) | Baseline, 6 weeks post-antibiotic therapy
Change in concentration of C-reactive protein (CRP) | Baseline, 6 weeks post-antibiotic therapy
Patient-Reported Outcomes Measurement Information System (PROMIS) - Global Health | Baseline, 6 weeks post-antibiotic therapy
  The PROMIS Global Health measure consists of 10 items designed to assess an individual's overall health status, encompassing physical, mental, and social well-being. Each item is scored on a Likert scale of 1-5. Scores are reported on a T-score metric, with a mean of 50 and a standard deviation of 10, meaning a score of 50 represents the average for the reference population. Higher scores indicate better health.
Hip Disability and Osteoarthritis Outcome Score for Joint Replacement (HOOS-JR) | Baseline, 6 weeks post-antibiotic therapy
  HOOS-JR contains 6 items from the original HOOS survey. Items are coded from 0 to 4, none to extreme, respectively. HOOS, JR is scored by summing the raw response (range 0-24) and then converting it to an interval score. The interval score ranges from 0-100, where 0 represents total hip disability and 100 represents perfect hip health.
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS-JR) | Baseline, 6 weeks post-antibiotic therapy
  KOOS-JR contains 7 items from the original KOOS survey. Items are coded from 0 to 4, none to extreme respectively. KOOS, JR is scored by summing the raw response (range 0-28) and then converting it to an interval score. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.

SECONDARY OUTCOMES:
Number of participants with medical complications from prosthetic joint infection (PJI) | 12 months post-surgery
  Outcome measure will be assessed using review of electronic medical record.
Number of participants with surgical complications from PJI | 12 months post-surgery
  Outcome measure will be assessed using review of electronic medical record.
Mortality from PJI | 12 months post-surgery
Digestion-associated Quality of Life Questionnaire (DQLQ) | 12 months post-surgery
  The DQLQ is a 9-items questionnaire assessing how digestive events and experiences affect mental well-being and physical ability. Participants respond based on how digestive events over the past seven days affected their quality of life using a 7-point frequency Likert scale (0 = never to 1 = always). Scores can range from 0 to 9; higher scores indicate a poorer digestion-associated quality of life.
The Short Health Scale for GI symptoms (SHS-GI) | 12 months post-surgery
  The SHS-GI is a 4-item questionnaire assessing the impact of gastrointestinal symptoms on quality of life, focusing on symptoms, social function, disease-related worry, and general well-being. Responses are graded on a 100-mm visual analog scale and maximum sum score for all items is 400, with higher values indicating worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ran Schwarzkopf, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: ran.schwarzkopf@nyulangone.org The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will need to execute a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: ran.schwarzkopf@nyulangone.org